CLINICAL TRIAL: NCT05535686
Title: Assessment of Adherence of Rheumatoid Arthritis Patients to Methotrexate and Its Effect on Quality of Life.
Brief Title: Methotrexate Adherence in Rheumatoid Arthritis Patients
Acronym: RA
Status: Completed | Type: Observational
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Abd El-Maboud, Marwa.M.Ad El-Maboud, Beni-Suef University
Other Study IDs: MTX in R.A
Record Dates: First submitted 2022-09-03; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rheumatoid Arthritis — Rheumatoid Arthritis Disease (R.A)

SUMMARY:
This study was conducted for assessment of adherence of Rheumatoid Arthritis patients to Methotrexate as a gold standard drug for treatment of R.A. Moreover, evaluating the effect of drug adherence to patient quality of life.

DETAILED DESCRIPTION:
Rheumatoid arthritis one of most common autoimmune diseases. characterized by numerous complications which may affect patient quality of life. Hence, this review aim to search the relation between patient"s drug adherence and clinical health outcome. our review utilizing survey as a tool to collect needed data from rheumatoid patients. survey consisted of number of questions , participants were required to answer these questions. participation to this questionnaire was optional.

ELIGIBILITY:
Inclusion Criteria:

1. The study was carried out among all RA patients (adults patients ≥ 18 years).
2. Patients not suffering from severe mental disorders.
3. Patients with a disease duration from (1-5) years.
4. Patients on MTX treatment from (1-5) years.
5. Patients taking MTX alone or in combination with other DMARDs.

Exclusion Criteria:

1. Patient who on MTX for more than 5 years
2. Patient who have complications like:-

   * History of liver or kidney disease
   * Diabetic patients
   * Hypertensive patients
   * Bone marrow hypoplasia
   * Leukopenia or significant anemia
   * Peptic ulcer or any GIT problems
   * Hereditary alopecia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The survey participants were adults diagnosed as RA patients in accordance to 2010 ACR/EULAR classification criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Rheumatoid Arthritis patient adherence to Methotrexate and its effect on quality of life | Baseline
  aim of this study was to measure Rheumatoid Arthritis patient adherence to MTX. A descriptive cross-sectional study was conducted on 300 RA patients administrating MTX for at least one year. Direct interview was used to complete the survey. The documented data were demographics (age, education , sex, work status). Patients' adherence to MTX as well as predictors for non-adherence.This investigational clinical study was conducted on RA outpatient clinic. Clinical parameters such as disease duration, duration on MTX therapy in years and current dose of MTX in milligrams per week were all documented.Structured questionnaire was designed to assessed the following areas: MTX side effects, patient adherence towards MTX, functional disability and patient awareness towards MTX. Patients were questioned about the prevalence of gastrointestinal adverse effects related to MTX. All data was collected from one direct interview with each RA patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Marwa, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No